CLINICAL TRIAL: NCT07225933
Title: A Retrospective, Multi-center Real-world Study of Steerable Ureteroscopic Renal Evacuation (SURE) Procedure With the CVAC® System
Acronym: REASON
Status: Active, not recruiting | Type: Observational
Sponsor: Calyxo, Inc. (Industry)
Collaborators: University of California, San Diego (Other); University of Alabama at Birmingham (Other); University of Texas Southwestern Medical Center (Other); OhioHealth Research Institute (Unknown); Feinstein Institute for Medical Research (Other); Summit Medical (Unknown); Western New York Urology Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: CP00005
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Urolithiasis; Kidney Stone; Kidney Stones
Keywords: SURE; FANS
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System: The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Interventions: Device: CVAC® SYSTEM
- FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS): FANS is designed to incorporate suction to facilitate stone fragment removal through its lumen and is used with a separate ureteroscope. FANS is fitted with a Y connector with a pressure control vent and connects to a standard vacuum device. A separate ureteroscope provides direct visualization and irrigation and a separate specimen collector captures stone debris.
  Interventions: Device: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS)

INTERVENTIONS:
Device: CVAC® SYSTEM — The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Other Names: SURE; CVAC
  Groups: Steerable Ureteroscopic Renal Evacuation (SURE) with CVAC System
Device: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS) — FANS is designed to incorporate suction to facilitate stone fragment removal through its lumen and is used with a separate ureteroscope. FANS is fitted with a Y connector with a pressure control vent and connects to a standard vacuum device. A separate ureteroscope provides direct visualization and irrigation and a separate specimen collector captures stone debris.
  Other Names: FANS; fURS
  Groups: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS)

SUMMARY:
This is a retrospective, multi-center collaboration to assess real-world outcomes of a novel steerable aspiration system, the CVAC® System ("CVAC"), and flexible and navigable suction ureteral access sheath (FANS) for the treatment of urinary stones.

DETAILED DESCRIPTION:
The objective of this study is observation of the safety and efficacy of subjects who underwent SURE procedure using the CVAC System or FANS for the removal of kidney stones in candidates for URS with laser lithotripsy. Efficacy will be observed by reviewing stone free status on standard of care post-procedure imaging. Safety will be observed by reviewing procedural information and if subjects had urologic events leading to Emergency Department (ED) visits, hospitalization, or retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that had SURE procedure with CVAC System performed in the retrospective cohort
* Subjects that had flexible URS (fURS) procedure with FANS performed in the retrospective cohort

Exclusion Criteria:

* For planned SURE procedures, the inability for CVAC to gain access required for treatment of kidney stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that are 18 or older that underwent the SURE procedure with the CVAC System or fURS with FANS in the retrospective cohort
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Stone free Status | Post-Operative up to 90 Days
  Completed by reviewing any available standard of care post-procedure imaging
Intra- & Post-Operative Complications | Intra- & Post-Operative up to 90 Days
  Completed by reviewing data available for intra- and post-op complications

CONTACTS AND LOCATIONS:
Overall Officials: Roger Sur, MD, Principal Investigator — UC San Diego
Locations (1):
- University of California San Diego (UCSD), La Jolla, California, United States